CLINICAL TRIAL: NCT02507011
Title: Beta-blockers in Pulmonary Arterial Hypertension - A Phase 2 Double-Blind, Placebo-Controlled, Crossover Study Evaluating the Efficacy, and Safety of Carvedilol for Right Ventricular Dysfunction in Pulmonary Arterial Hypertension
Brief Title: Beta-blockers in Pulmonary Arterial Hypertension
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1504M69361
Record Dates: First submitted 2015-07-22; First posted 2015-07-23 (Estimated); Results first posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-05

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Carvedilol; Adrenergic beta-Antagonists

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Carvedilol First (Experimental): Crossover Design: Participants receive Carvedilol first and placebo second
  Interventions: Drug: Carvedilol; Drug: Placebo
- Placebo First (Placebo Comparator): Crossover Design: Participants receive placebo first and Carvedilol second
  Interventions: Drug: Carvedilol; Drug: Placebo

INTERVENTIONS:
Drug: Carvedilol — Beta-adrenergic receptor blocker
  Other Names: Beta-blockers
Drug: Placebo — Placebo

SUMMARY:
The investigators will conduct a, randomized, phase 2, placebo-controlled, double-blinded, crossover trial of carvedilol in 26 PAH patients with World Health Organization functional class II or III symptoms and RV ejection fraction (EF) < 45% for 6 months.

DETAILED DESCRIPTION:
Adult PAH patients on a stable dose of an approved PAH medication will undergo the following baseline assessments: cardiac magnetic resonance imaging (MRI), right heart catheterization (RHC), echocardiogram, 6-minute walk test (6-MWT), plasma NT-ProBNP (biomarkers of RV function) and serum catecholamine (measure of sympathetic activation), and quality of life. Patients will be randomized to carvedilol (3.125 mg bid and escalated to 9.375 mg bid, as tolerated, over 3 months) or placebo in a 1:1 fashion. After 6 months, testing is repeated and patients are crossed over to the alternate treatment. Testing is repeated at the end of the study (month 13).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* WHO category 1 pulmonary arterial hypertension (Nice 2013)
* WHO functional class II-III
* RVEF by cardiac MRI < 45%
* Stable on PAH-specific therapy as defined by no change in PAH-specific treatment and functional class in the past 3 months. Patient can be on either mono or combination PAH-specific therapy

Exclusion Criteria:

* Subjects will be excluded from participation in the study if any of the following conditions exist:
* Significant persistent bradycardia (resting heart rate < 60 bpm) without a permanent pacemaker
* Second or third degree AV block without a permanent pacemaker
* Significant sinus tachycardia (resting heart rate > 110 bpm)
* Use of anti-arrhythmic drugs
* Hypotension defined as systolic blood pressure < 100 mmHg at the time of enrollment
* Significant illness in the past 30 days requiring hospitalization
* Acute decompensated right heart failure within past 30 days
* Known allergy or intolerance to carvedilol or other β blockers
* Cardiac index < 2 l/min/m2 or right atrial pressure > 15 mm Hg by right heart catheterization within last 3 months
* Asthma
* Positive pregnancy test in patients of child bearing-potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-01-31 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thenappan Thenappan, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Medical Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Carvedilol First, Then Placebo: Participants in this arm received Carvedilol first
- Placebo First, Then Carvedilol: Participants in this arm received placebo first
Period: First Intervention
Arm/Group | Carvedilol First, Then Placebo | Placebo First, Then Carvedilol
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Carvedilol First, Then Placebo | Placebo First, Then Carvedilol
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Crossover Design: All participants pooled at baseline
Arm/Group | All Participants
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Right Ventricular Ejection Fraction as Measured by Cardiac MRI
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percent
Groups:
- Carvedilol: Beta Blocker
  Carvedilol: Beta-adrenergic receptor blocker
  Placebo: Placebo
- Placebo: General Placebo
  Carvedilol: Beta-adrenergic receptor blocker
  Placebo: Placebo
Arm/Group | Carvedilol | Placebo
Number analyzed (Participants) | 2 | 2
percent | 10 (4) | 2.5 (2)

ADVERSE EVENTS:
Time Frame: 13 months
Arm/Group | Carvedilol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2 | 1/2
Other Adverse Events (participants affected / at risk) | 1/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carvedilol (N=2) | Placebo (N=2)
HF Exaceberation/Electrolyte Imbalance (General disorders) | 1 (3) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carvedilol (N=2) | Placebo (N=2)
Fatigue (General disorders) | 1 (1) | 1 (1)
Hypotension (General disorders) | 1 (1) | 0 (0)
Fluid Retention (General disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (2)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2017-10-12): https://cdn.clinicaltrials.gov/large-docs/11/NCT02507011/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-10-12): https://cdn.clinicaltrials.gov/large-docs/11/NCT02507011/Prot_SAP_001.pdf